CLINICAL TRIAL: NCT03811379
Title: Phase II Clinical Trial of Toripalimab (JS001), a Recombinant Humanized Anti-PD-1 Monoclonal PD1 Antibody, as Monotherapy for Patients With Small Cell Esophageal Carcinoma Who Failed Chemotherapy
Brief Title: Toripalimab as Monotherapy for Patients With Small Cell Carcinoma of Esophagus Who Failed Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ruihua Xu, President and professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PD-1/SCCE
Record Dates: First submitted 2019-01-17; First posted 2019-01-22 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Small Cell Carcinoma of Esophagus; Advanced Cancer
Keywords: Immunotherapy
MeSH Terms: interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toripalimab (Experimental): Toripalimab, 240mg, every 3 weeks until disease progress or intolerable toxicity
  Interventions: Drug: Toripalimab

INTERVENTIONS:
Drug: Toripalimab — Drug: Toripalimab, 240mg, every 3 weeks until disease progress or intolerable toxicity

SUMMARY:
To evaluate the anti-tumor activity, safety and tolerance of toripalimab as monotherapy for patients with small cell esophageal cancer (SCCE), and to explore the potential biomarkers for this treatment.

DETAILED DESCRIPTION:
For the first time in the world, the investigators revealed the genomic characteristics of SCCE and constructed a complete genomic profile of SCCE. The analysis of transcriptome data showed that the number of effector T cells in SCCE immune microenvironment was significantly higher than that of other cancers, and NK cells were relatively high. Macrophages in SCCE mainly showed M2-like phenotype and maintained at a relatively high level, suggesting the possibility of immunotherapy in SCCE treatment. Therefore, the purpose of this study is to clarify the efficacy of PD-1 antibody in the treatment of patients with SCCE who failed chemotherapy, so as to provide a basis for further large-scale clinical research.

ELIGIBILITY:
Inclusion Criteria:

1. Full understanding of the study and voluntary signing of informed consent
2. Histologically and/or cytologically confirmed advanced and/or metastatic small cell carcinoma of the esophagus who failed previous first-line or more lines of chemotherapy or the disease recurs within six months after the adjuvant or neoadjuvant therapy
3. At least one measurable lesion (according to RECIST 1.1) Note: Lesions previously treated with radiotherapy should not be considered as target lesions unless there is a definite progression after radiotherapy.
4. Agree to provide previously stored specimens of tumor tissue or to perform biopsy to collect tumor tissue for PD-L1 IHC detection.
5. The age ranges from 18 to 75 years with no gender limitation.
6. ECOG: 0-1
7. Expected survival ≧ 3 months
8. Laboratory tests within 7 days before admission must meet the following criteria: A. Neutrophils≧1.5 *109/L; B. Platelet ≧ 75 *109/L; C. Hemoglobin≧90g/L (no infusion of concentrated red blood cells within 2 weeks); D. Serum creatinine≦1.5 * ULN, or creatinine clearance rate > 50 mL/min; E. Serum total bilirubin ≦ 1.5 *ULN (Gilbert syndrome subjects allowed total bilirubin ≦ 3 *ULN); F. AST and ALT ≦ 2.5 *ULN, while ALT and AST were less than 5 *ULN in subjects with liver metastasis.
9. Within 21 days before admission, women of childbearing age must confirm that the serum pregnancy test is negative and agree to use effective contraceptive measures during the study period and within 28 days after the last administration. Female reproductive age in this program is defined as sexually mature women: 1) without hysterectomy or bilateral ovariectomy, 2) natural menopause without continuous 24 months (menopause after cancer treatment does not exclude fertility) (Menstruation occurs at any time during the previous 24 consecutive months).

Exclusion Criteria:

1. known to be allergic to citric acid monohydrate, sodium citrate dihydrate, mannitol and polysorbide (components of the test drug).
2. Within the first four weeks of admission, patients received anti-tumor cytotoxic drugs, biological drugs (such as monoclonal antibodies), immunotherapy (such as interleukin-2 or interferon), or other research drugs.
3. Tyrosine kinase inhibitors were administered within 2 weeks before admission.
4. Radiotherapy or radiopharmacotherapy were given within 4 weeks or 8 weeks before admission, except local palliative radiotherapy for bone metastases.
5. Major surgical operations were performed or not fully recovered from previous operations within the first four weeks of enrollment (the definition of major surgical operations refers to the 3-and 4-level operations stipulated in the Regulations on the Clinical Application of Medical Technologies, which were implemented on 1 May 2009).
6. The toxicity of previous antineoplastic therapies has not been restored to CTCAE 0-1, except for the following cases:

   A alopecia; B pigmentation; C Peripheral neurotoxicity has been restored to < CTCAE level 2. D The long-term toxicity caused by radiotherapy can not be restored by the judgement of the researchers.
7. Subjects with clinical symptoms of central nervous system metastasis (e.g. brain edema, requiring hormone intervention, or progression of brain metastasis) and/or cancerous meningitis. Subjects who had previously received brain or meningeal metastasis therapy, such as clinical stability maintained for at least two months, and who had stopped systemic sex hormone therapy (prednisone or other therapeutic hormones at doses greater than 10 mg/day) for more than four weeks could be included.
8. Other malignant tumors (besides skin basal cell carcinoma, breast/cervical carcinoma in situ, and other malignancies that have not been treated and effectively controlled in the past five years) have been or are currently co-existing with other malignant tumors.
9. Subjects had any history of active autoimmune diseases or autoimmune diseases (including, but not limited to, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, nephritis, hyperthyroidism, hypothyroidism); subjects with vitiligo or childhood asthma had been completely alleviated; subjects without any intervention after adulthood could be included in the study; Asthma, which requires medical intervention with bronchodilators, cannot be included.
10. Anti-PD-1 antibody, anti-PD-L1 antibody, anti-PD-L2 antibody or anti-CTLA-4 antibody (or any other antibody acting on T cell co-stimulation or checkpoint pathway) have been used in the past.
11. Subjects with active pulmonary tuberculosis (TB) are receiving anti-tuberculosis treatment or anti-tuberculosis treatment within one year before screening.
12. Complications of corticosteroids requiring long-term use of immunosuppressive drugs or systemic or local use of prednisone or other therapeutic hormones with an immunosuppressive dose of more than 10 mg/day.
13. Any anti-infective vaccines (such as influenza vaccine, varicella vaccine, etc.) were inoculated within 4 weeks before admission.
14. Pregnant or lactating women.
15. HIV positive.
16. HBsAg positive and HBV DNA copy number positive (quantitative detection ≧ 1000 cps/ml).
17. Blood screening for chronic hepatitis C is positive (HCV antibody is positive).
18. Researchers believe that it may affect program compliance, or the signing of informed consent (ICF), or any other disease or condition of clinical significance that is not suitable for this clinical trial.
19. Heart clinical symptoms or diseases that have not been well controlled, such as:

(1) heart failure above NYHA Level 2 (2) unstable angina pectoris (3) myocardial infarction within 1 year (4) clinically significant supraventricular or ventricular arrhythmias need treatment or intervention;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2018-11-21 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rates (ORR) | up to two year
  the ratio of patients who are evaluated as CR or PR

SECONDARY OUTCOMES:
Progression free survival (PFS) | up to two year
  defined as the time from the first dose of study treatment to disease progression
Overall Survival (OS) | up to two year
  defined as the period from the first dose of study treatment to loss of follow-up or death
Duration of remission (DOR) | up to two year
  Defined as the time between the first assessment of a tumor as PR or CR and the first assessment as PD or any cause of death
Disease Control Rate (DCR) | up to two year
  It is defined as the proportion of patients whose tumors shrink or remain stable for a certain period of time, including CR, PR and SD.
Adverse Events (AEs) | up to two year
  All treatment-related adverse events (AEs) were categorized according to the National Cancer Institute's Common Terminology Criteria for Adverse Events.

CONTACTS AND LOCATIONS:
Overall Officials: Rui-hua Xu, MD, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Cancer center of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided